CLINICAL TRIAL: NCT07294924
Title: PREDICT-ACC: Prediction of REsponse to Depression Interventions (Accelerated rTMS) Using Clinical and TD-fNIRS Measurements
Brief Title: Prediction of REsponse to Depression Interventions (Accelerated rTMS) Using Clinical and TD-fNIRS Measurements
Acronym: PREDICT-ACC
Status: Recruiting | Type: Observational
Sponsor: Kernel (Industry)
Collaborators: Acacia Clinics (Unknown)
Responsible Party: Sponsor
Other Study IDs: KER2025-1-PREDICT-ACC
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder (MDD); fNIRS
Keywords: Accelerated TMS; Healthy Controls; Observational; Longitudinal; Neuroimaging
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Accelerated TMS Cohort: Participants who have previously been diagnosed with MDD and have elected to undergo accelerated TMS to treat their depression at a participating clinic will be enrolled in the study.
  Interventions: Other: fNIRS measurement
- Healthy Controls Cohort: Participants with no diagnosis of depression and no depression-related treatment within the past year will be enrolled as the control group.
  Interventions: Other: fNIRS measurement

INTERVENTIONS:
Other: fNIRS measurement — Kernel Flow is a non-invasive neuroimaging device that uses time-domain functional near-infrared spectroscopy (TD-fNIRS) to measure changes in cortical hemodynamics associated with brain activity.
  Other Names: Kernel Flow

SUMMARY:
This observational, longitudinal, multi-cohort study aims to evaluate functional brain activity in adults undergoing treatment for Major Depressive Disorder (MDD) at participating clinical sites. A separate cohort of healthy adults will be enrolled as a control group. All data collected in this study are for research purposes only and will not influence clinical decision-making or treatment plans.

This study will use TD-fNIRS to measure hemodynamic brain responses at rest and/or during tasks in patients receiving accelerated transcranial magnetic stimulation (TMS). Imaging will occur at multiple timepoints (pre-treatment, post-treatment, and follow-ups). Healthy control participants will complete similar measurements at one visit, with the option for a follow-up visit. The primary objectives are to assess feasibility, characterize brain activity patterns, and explore potential biomarkers associated with treatment response.

ELIGIBILITY:
Inclusion Criteria for:

Accelerated TMS cohort

* Adults aged 18-75 at the time of enrollment
* Primary diagnosis of MDD as defined by the DSM-5
* Determined by the clinic to be eligible for accelerated rTMS treatment and agrees to receive accelerated rTMS treatment
* Agrees to start accelerated rTMS treatment in conjunction with study participation to capture baseline measurements
* Has not received rTMS treatment in the past 1 month
* Has not received SPRAVATO treatment in the past 1 month
* Can speak and understand English
* Ability to provide informed consent

Healthy controls cohort

* Adults aged 18-75 at time of enrollment
* Can speak and understand English
* Ability to provide informed consent

Exclusion Criteria for:

All cohorts

* Pregnant or may become pregnant during the treatment course
* Unable or unwilling to wear the fNIRS headset
* Has had electroconvulsive therapy (ECT) in the past 3 months
* Major medical illnesses including neurological and psychiatric conditions such as Alzheimer's disease, Parkinson's disease, multiple sclerosis, epilepsy, schizophrenia, or stroke.
* Any other clinically significant medical condition that in the opinion of the clinician or study team, could affect patient safety, wellbeing, or the participant's ability to comply with study procedures.
* Not an appropriate candidate for the study based on the discretion of the study investigator(s).

Healthy controls cohort only

* Clinical diagnosis of depression in the past year
* Undergoing any treatments for depression in the past year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes two cohorts of adults aged 18-75: (1) participants with a primary diagnosis of Major Depressive Disorder (MDD) who are eligible for and agree to undergo accelerated rTMS treatment, and (2) healthy control participants with no depression diagnosis or depression-related treatment in the past year. All participants must be able to provide informed consent, speak English, and meet general safety and eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
TD-fNIRS Biomarkers of Treatment Response and Group Differences | Up to 20 minutes during each study visit
  To gather hemodynamic data with TD-fNIRS and develop biomarkers of depression treatment response and group differences between patients and controls. Candidate markers to relate to clinician assessments are:
  1. Local changes in neural activity during Resting State and Task;
  2. Functional Connectivity during Resting State and Task;
  3. Patterns of Hemodynamic Responses During Emotional, and/or Verbal Fluency Tasks

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Perdue, PhD, Principal Investigator — Kernel
Locations (2):
- United States (2):
  - Kernel, Los Angeles, California
  - Acacia Clinics, Sunnyvale, California

IPD SHARING:
Plan to Share IPD: Undecided